CLINICAL TRIAL: NCT05918887
Title: Feasibility and Acceptability of Switching to E-cigarettes Among Cigarette Smokers Engaged in Substance Use Disorder Treatment
Brief Title: Feasibility and Acceptability of Switching to E-cigarettes Among Cigarette Smokers Engaged in SUD Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Principal Investigator, Jennifer Pearson, Associate Professor, University of Nevada, Reno
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2040809
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Dependence Caused by Cigarettes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- E-cigarette arm (Experimental): Participants will receive the commercially available NJOY ACE e-cigarette, nicotine pods (2 of each available flavor, for a total of 4 pods), and tailored instructions to switch. Participants will use the ACE ad libitum for 14 days, reporting their cigarette use, e-cigarette use, mood, and nicotine crazing every day via text message surveys.
  Interventions: Device: NJOY ACE commercial e-cigarette

INTERVENTIONS:
Device: NJOY ACE commercial e-cigarette — The NJOY ACE is the commercial version of the Standardized Research E-Cigarette (SREC), which was developed by NIDA with NJOY for research purposes.
  Nicotine pods:
  * Sealed, pre-filled, non-refillable
  * 1.9 mL e-liquid with 5% w/w nicotine
  * Approx 300 (280-330) puffs/pod
  Nicotine liquid characteristics:
  * Volume of liquid per pod 1.9 mL
  * Active (nicotine USP 5% wt/wt)
  * Propylene Glycol USP & Vegetable Glycerin USP - PG/VG Ratio 0.77
  * Lactic Acid USP
  Battery characteristics:
  * USB Rechargeable
  * Storage Capacity ~ 400 mAh
  * Approx 200 (3s) puffs / charge
  * 300 charge cycles to > 80% initial capacity
  * Time to full charge 75 - 85 min
  * Voltage / Temperature settings not user adjustable

SUMMARY:
The purpose of the proposed study is to examine the feasibility of integrating a smoking harm reduction program featuring provision of e-cigarettes and tailored instructions to switch into an existing substance use disorder treatment program. This longitudinal study includes three weeks of micro-surveys delivered via text messages to evaluate the intervention's feasibility and acceptability, gather initial effectiveness data, and understand participants' lived experience of smoking and vaping while engaged in substance use disorder treatment.

DETAILED DESCRIPTION:
The purpose of this study is to examine the feasibility of integrating a smoking harm reduction program featuring provision of e-cigarettes and tailored instructions to switch into an existing substance use disorder treatment program.

The proposed longitudinal study will include three weeks of micro-surveys delivered via text messages (called ecological momentary assessments, or EMA) to evaluate the intervention's feasibility and acceptability, gather initial effectiveness data, and understand participants' lived experience of smoking and vaping while engaged in substance use disorder treatment. As people gain access to substance use disorder treatment and the acute risk of death due to overdose diminishes, there is a significant need for data-driven, novel, and scalable smoking harm reduction approaches that meet people in recovery "where they are" and help them live longer, healthier lives by either significantly reducing their smoking frequency or switching completely to a much lower harm nicotine product.

Up to 30 daily cigarette smokers who are engaged in a substance use disorder treatment program and are not interested in quitting nicotine use but are interested in reducing the harm from smoking will be enrolled in the study. Aims include:

Aim 1. Examine the feasibility (e.g., enrollment, attrition), acceptability (e.g., e-cigarette use rates, user experience), and effectiveness (e.g., % who reduced smoking by at least 50% in Week 3 vs. Week 1; % who switched completely at Week 3) of the intervention on cigarette smoking among people engaged in substance use disorder treatment. It is anticipated that of the 30 people enrolled, 20 will complete the protocol. In Week 1, participants will report their usual smoking to establish baseline behavior. In Week 2, participants will be provided with an e-cigarette, nicotine liquid, and instructions to switch developed in Aim 1. In Week 3, participants' nicotine liquid supply will be replenished, and data collection will continue.

Aim 2. Describe participants' understanding of the meaning and utility of cigarettes and e-cigarettes in their lives. Up to 20 participants will take part in a semi-structured interview at the end of Week 3. Interviews will focus on their experience trying to switch while engaged in substance use disorder treatment and how their cognitions, expectancies, social relationships, and norms evolved over the 2 weeks of e-cigarette use. Qualitative data will complement quantitative data, adding participants' understanding of the "why" driving their behavior to the "what" captured with EMA, and will identify opportunities to improve the intervention and identify blind spots in our assessments for the main study. In-depth interviews also facilitate investigation of exploratory hypotheses that arise during data collection, suggesting additional areas of inquiry for a subsequent R01 proposal.

ELIGIBILITY:
Inclusion Criteria:

1. currently engaged in outpatient treatment the Mathewson Institute (medication, behavioral, or combination treatment) or other local treatment center
2. aged 21+
3. interested in switching from cigarettes to e-cigarettes, assessed by the item "Are you interested in replacing some or all of your cigarettes with e-cigarettes?"
4. has a cellphone with an unlimited text message plan
5. has had the same phone number for at least 1 month
6. uses text messages at least once a week
7. self-reports daily smoking
8. records an exhaled air carbon monoxide (CO) level >6ppm at baseline study visit
9. has the capacity to understand the participant materials and follow the study procedures (e.g. sufficient English language ability).

Exclusion Criteria:

Individuals who meet any the following criteria will not be enrolled in this study:

1. have used an e-cigarette to quit smoking in the past month
2. are currently pregnant or breast-feeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Change in average number of cigarettes consumed - Week 2 vs. Week 1 | Week 2 vs. Week 1
  Change in average cigarette consumption per day as a function of daily e-cigarette use
Change in average number of cigarettes consumed - Week 3 vs. Week 1 | Week 3 vs. Week 1
  Change in average cigarette consumption per day as a function of daily e-cigarette use

SECONDARY OUTCOMES:
Recruitment feasibility | Week 1
  50% of people who are screened for the study who are eligible and consent to participate in the study at Study Visit 1
Attrition feasibility | Through study completion, up to Week 4
  66.6% of consented participants will complete the study
Adherence fidelity | Weeks 2 and 3
  80% of people who report using the e-cigarette at least once a day in Weeks 2 and 3
EMA scheduled prompt feasibility | Weeks 1-3
  80% of people who complete at least 1 scheduled prompt a day
EMA random prompt feasibility | Weeks 1-3
  80% of people who complete at least 1 random prompt a day

OTHER OUTCOMES:
Smoking reduction | Week 3 vs. Week 1
  Percent of participants who reduced their smoking by at least 50%
Complete switching to e-cigarettes | Week 3
  Percent of participants who completely switched to e-cigarettes by the end of Week 3

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada, Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No